CLINICAL TRIAL: NCT04224402
Title: Phase 2 Trial to Investigate the Efficacy and Safety of mFOLFIRINOX as Postoperative Chemotherapy for Pancreatic Cancer in Chinese Patients.
Brief Title: Efficacy and Safety of mFOLFIRINOX as Postoperative Chemotherapy for Pancreatic Cancer in Chinese Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOLFIRINOX-PC-Adjuvant
Record Dates: First submitted 2019-12-06; First posted 2020-01-13 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Cancer Resectable

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mFOLFIRINOX (Other): Patients will receive mFOLFIRINOX every 2 weeks: Oxaliplatin 65 mg/m2 IV over 3 hours on Day 1; Irinotecan 150 mg/m2 IV over 90 minutes on Day 1; Leucovorin(l-LV) 200 mg/m2 IV over 2 hours on Day 1; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion
  Interventions: Drug: mFOLFORINOX

INTERVENTIONS:
Drug: mFOLFORINOX — Patients will receive mFOLFIRINOX every 2 weeks: Oxaliplatin 65 mg/m2 IV over 3 hours on Day 1; Irinotecan 150 mg/m2 IV over 90 minutes on Day 1; Leucovorin(l-LV) 200 mg/m2 IV over 2 hours on Day 1; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion.

SUMMARY:
This prospective and open-label study evaluates the efficacy and safety of mFOLFIRINOX as postoperative chemotherapy in treating Chinese patients with pancreatic cancer after R0/R1 resection.

DETAILED DESCRIPTION:
The patients will be treated with systemic FOLFIRINOX chemotherapy of adjusted dosage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should be voluntary to the trial and provide with signed informed consent.
2. Histologically confirmed diagnosis of pancreatic cancer
3. Male or female, Age: 18-79 years old.
4. No recurrence or metastasis was observed from a follow-up of 4 to 8 weeks by CT scan after radical surgery.
5. the value of Carbohydrate Antigen19-9(CA19-9) < 180U/mL within 12 weeks after surgery.
6. No previous chemotherapy
7. Eastern Cooperative Oncology Group(ECOG) performance status of 0-1
8. normal function of organ system including the followings.

   * No hematologic dysfunction(Platelets ≥90×10^9/L; Neutrophil ≥2×109/L;Hemoglobin ≥90g/L).
   * Serum bilirubin ≤ 1.2 × upper limits of normal(ULN); aminotransferase ≤ 5 × ULN.
   * Serum creatinine ≤ 1.25× ULN, or creatinine clearance rate(CCR) ≥60mL/min(calculated by Cockcroft-Gault formula).
9. ECOG scored as 0-1.
10. Life expectancy > 3 months.

Exclusion Criteria:

1. Patient is concurrently using other antineoplastic agent.
2. Known severe hypersensitivity to drugs in the regimen.
3. Patient has a concurrent malignancy or has a malignancy within 5 years of study enrollment(with the exception of nonmelanoma skin cancer or cervical carcinoma in situ).
4. Evidence of serious heart disease, including recorded history of congestive heart-failure, uncontrolled serious arrhythmia, angina that needs treatment of drugs, clinical diagnosed cardiac valve disease, history of serious myocardial infarction and intractable hypertension.
5. Evidence of chronic diarrhea(≥4 times/day) or renal dysfunction.
6. Evidence of active infection or active epidemic disease.
7. Psychiatric illness that would prevent the patient from giving informed consent
8. Pregnant or lactating women.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Regression Free Survival | Up to 24 months
  defined as the period from the date of resection to tumor relapse caused by any reason

SECONDARY OUTCOMES:
Overall Survival | Up to 24 months
  the duration from enrollment to the patient's death (all causes)

OTHER OUTCOMES:
adverse events and severe adverse events | Up to 12 weeks
  number of patients with adverse events and severity according to NCI Common Toxicity Criteria(CTC) 3.0
EORTC Quality of Life Questionnaire(QLQ)-C30 | Up to 24 weeks
  Quality of life will be assessed at each study using EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Yu-hong Li, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China